CLINICAL TRIAL: NCT05621876
Title: Evaluation of an IgG Deficiency Rapid Screening Test (RDT) With Human Capillary Samples: A Protocol to Generate RDT Performance Data in Primary Immunodeficiency Patients (PID)
Brief Title: Evaluation of an IgG Deficiency Rapid Screening Test: A Performance Study With Primary Immunodeficiency (PID) Patients in Tunisia
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Institut Pasteur de Tunis (Other); Centre National de Greffe de Moelle Osseuse (Other Government)
Responsible Party: Principal Investigator, Megan Parker, Senior Program Officer, PATH
Other Study IDs: 1923231
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Primary Immunodeficiency Diseases
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will be retaining small amounts of plasma to be held at IPT in Tunisia for future testing. We are asking study participants if they want to contribute samples to the biorepository. No samples will be obtained without their consent. These samples will be de-identified, and only be labelled with the type of PID the child experiences. There are 400 different types of primary immunodeficiencies and we are trying to improve low-cost diagnostics to detect all types to detect low IgG individuals to prevent the spread of polio from the polio vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: IgG deficiency rapid screening test — We will be testing patients who have already been diagnossed iwth primary immunodeficiency (PID) disease. there are 400 types of PID. We will test their blood before they receive antibody transfusion to evaluate the accuracy of our new screening test. We are trying to develop easy to use, low-cost screening tests for doctors to use with patients to detect those with low IgG levels before they are given the oral polio vaccine. These patients must be prioritized for intramuscular injections of a polio vaccine to prevent potential spread of wild type polio.

SUMMARY:
To evaluate the usability and utility of the device, % agreement between the PID-RDT and the referent assay (serum/plasma), and % agreement between capillary blood and venous blood samples using the PID-RDT within confirmed PID patients prior to receipt of their monthly IV-Ig treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be 6 months of age.
* The types of PID presenting for IV-Ig therapy will include Evaluation of PID RDT with human capillary blood (version 1.0) | 8agammaglobulinemia (AG), hypogammaglobulinemia (HAG), common variable immunodeficiency (CVID), and hyper IgM syndrome (HIGM).

Exclusion Criteria:

-

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: PID patients prior to receiving IV-Ig treatment infusions for the first time or during follow-up at the NBMT center in Tunis. The day of their monthly infusion, they are expected to have the lowest residual IgG level. These patients have previously been identified with AG, HAG, CVID and HIGM and this is why they are receiving IV-Ig therapy at NBMT. Patients will be 6 months of age or older and the patient or guardian must give consent for participation.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
To evaluateusability among end users of the PID rapid screening tests using capillary blood samples obtained from PID patients, prior to receipt of IV-Ig treatment. | 3 month
  - Did the test run correctly when following the IFU?
  •Was the end user (nurse) able to interpret a test result for the patient from the investigational PID RDT (positive, negative) with valid control using a patient's capillary finger prick sample?
To evaluate % agreement between the PID RDT(using capillary blood)and the referent test (serum/plasma). | 3 months
  What is the % agreement between the PID RDT run on capillary blood (Capillary Test A) and the referent assay run on plasma/serum?

SECONDARY OUTCOMES:
To determinethe utility of the PID RDTwith PID patients. | 3 months
  Can the investigational PID RDT be used with a finger prick (capillary) blood sample among study participants?
  * Was the finger prick blood sample successfully collected from the finger and transferred to the PID RDT?•Did the test run complete and give a valid result when run according to instructions?
  * Could a result be interpreted from the PID RDT?
To determine% agreement between capillary and venous blood samples using the PID RDT | 3 months
  What is the % agreement between fresh capillary blood and fresh venous blood using the PID RDT?

CONTACTS AND LOCATIONS:
Locations (1):
- National Bone Marrow Transplant center, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
Knowledge gained from this study may benefit society by providing information on the diagnostic accuracy of the first PID RDT. Data obtained from this study will be made available to the test manufacturer to support their product dossier, and ultimately to provide countries still working to eradicate polio with quality-assured PID RDTs with analytical and clinical performance beyond that provided by the Jeffrey Modell warning signs.